CLINICAL TRIAL: NCT06399809
Title: Fisetin to Reduce Senescence and Mobility Impairment in Peripheral Artery Disease: the FIRST Pilot Randomized Trial
Brief Title: Fisetin to Reduce Senescence and Mobility Impairment in PAD
Acronym: FIRST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00217306
Record Dates: First submitted 2023-10-28; First posted 2024-05-06 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease; Aging; Peripheral Vascular Diseases; Walking, Difficulty; Claudication
Keywords: Fisetin
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Mobility Limitation; Intermittent Claudication | interventions — fisetin

STUDY DESIGN:
Intervention Model Description: To achieve the trial's specific aims, the investigators will randomize 34 participants age 50 and older with PAD to one of two groups: Fisetin vs placebo. Participants will be followed for four months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double blinded study where both the participant and the investigators collecting data will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fisetin (Experimental): Sharp Clinical Services will provide fisetin (100 mg capsules). Randomized participants will receive fisetin 20 mgs/kg once daily for two days, followed by 12 days without therapy. Fisetin will be dosed in 100 mg tablets. Dosing will be rounded to the nearest 100 mg. For example, a 73 kg participant with a dose of 1,460 mg (i.e.73 kg x 20 mg) receives 1,500 mgs daily (i.e. 15 x 100 mg capsules) for two days every 14 days.
  Interventions: Drug: Fisetin
- Placebo (Placebo Comparator): Sharp Clinical Services will provide placebo (100 mg capsules). Randomized participants will receive placebo 20 mgs/kg once daily for two days, followed by 12 days without therapy. Placebo will be dosed in 100 mg tablets. Dosing will be rounded to the nearest 100 mg. For example, a 73 kg participant with a dose of 1,460 mg (i.e.73 kg x 20 mg) receives 1,500 mgs daily (i.e. 15 x 100 mg capsules) for two days every 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin — Fisetin is a flavanol, present in strawberries, apples, and persimmons, that destroys senescent cells (i.e. a senolytic therapy). Of three senolytic therapies being tested in clinical trials, fisetin has the best safety profile.
  Arms: Fisetin
Drug: Placebo — The placebo will be matched to the Fisetin intervention
  Arms: Placebo

SUMMARY:
The investigators propose a pilot randomized trial to gather preliminary data to test the hypothesis that Fisetin will reduce abundance of senescent cells in blood, skeletal muscle, and both subcutaneous and inter muscular adipose tissue and improve 6-minute walk distance in 34 people with peripheral artery disease (PAD). the investigators will determine whether greater declines in abundance of cells with senescent markers are associated with greater improvement in 6-minute walk distance in people with peripheral artery disease. In exploratory analyses, the investigators will assess whether Fisetin reduces interleukin-6 (IL-6) and novel senescent markers in adipose tissue, muscle, and/or blood.

DETAILED DESCRIPTION:
Fisetin is a flavanol, present in strawberries, apples, and persimmons, that destroys senescent cells (i.e. a senolytic therapy). Of three senolytic therapies being tested in clinical trials, Fisetin has the best safety profile. Hence, the investigators propose a pilot randomized trial to gather preliminary data to test the hypothesis that Fisetin will reduce abundance of senescent cells in blood, skeletal muscle, and both subcutaneous and inter muscular adipose tissue and improve 6-minute walk distance in 34 people with PAD. The investigators will determine whether greater declines in abundance of cells with senescent markers are associated with greater improvement in 6-minute walk distance in people with PAD. In exploratory analyses, the investigators will assess whether Fisetin reduces IL-6 and novel senescent markers in adipose tissue, muscle, and/or blood.

To achieve the trial's specific aims, investigators will randomize 34 participants age 50 and older with PAD to one of two groups: Fisetin vs placebo. Participants will be followed for four months.

ELIGIBILITY:
Inclusion Criteria:

First, all participants will be age 50 and older. Second, all participants will have PAD. PAD will be defined as:

1. An ankle brachial index (ABI) less than or equal to 0.90 at baseline.
2. Vascular lab evidence of PAD (such as a toe brachial pressure less than or equal to 0.70 or an ankle brachial index less than or equal to 0.90), or angiographic evidence of PAD defined as at least 70% stenosis of an artery supplying the lower extremities.
3. An ABI of greater than 0.90 and less than or equal to 1.00 who experience a 20% or greater drop in ABI in either leg after the heel-rise test will also be included.

Exclusion Criteria:

1. Above- or below-knee amputation
2. Critical limb ischemia defined as an ABI less than 0.40 with signs or symptoms of critical limb ischemia
3. Wheelchair confinement or requiring a walker to ambulate
4. Walking is limited by a symptom other than PAD
5. Current foot ulcer on bottom of foot
6. Failure to successfully complete the study run-in
7. Planned major surgery, coronary or leg revascularization during the next five months
8. Major surgery, coronary or leg revascularization or major cardiovascular event in the previous three months
9. Major medical illness including lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who require oxygen only at night may still qualify.]
10. Mini-Mental Status Examination (MMSE) score less than 23
11. Allergy to fisetin
12. Currently taking fisetin or has taken fisetin in previous three months
13. Non-English speaking
14. Current participation in or completion of a clinical trial intervention in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a clinical trial (other than stem cell or gene therapy), participants will be eligible after the final study intervention as long as at least three months have passed since the final intervention of the trial.]
15. Visual impairment that limits walking ability.
16. Six-minute walk distance of less than 500 feet or greater than1600 feet.
17. Participation in a supervised treadmill exercise program in previous three months.
18. Participants may be excluded if they are unwilling to undergo a fat biopsy. However, if investigators find recruitment significantly slows due to this exclusion, participants may still be able to participate in the trial if they refuse the fat biopsy.
19. Women who are not menopausal will be excluded. Menopause is defined as absence of a menstrual period in the past 12 months.
20. People with a bilirubin above 2.2 mg/dl, with serum aspartate transaminase (AST) or alanine aminotransferase (ALT) more than four times the upper limit of normal.
21. Hemoglobin less than 7.0 g/dl, white blood count less than 2,000/mm3, white blood count greater than 20,000/mm3, platelet count less than 40,000/uL.
22. Estimated glomerular filtration rate (eGFR) less than 25 ml/min/1.73 m2
23. HemoglobinA1C great than 10 as a marker of poor diabetes control.
24. People who are Human Immunodeficiency Virus positive (HIV+) and people with active hepatitis B or active hepatitis C infections who do not have a low viral load.
25. People taking warfarin and other sensitive substrates of CYP2C9, CYP2C19, or CYP1A2 that have a narrow therapeutic window will be excluded, unless the drug can be held for at least two days prior to the first day of each study drug administration and can continue to be held for ten hours after the second dose of study drug administration for each of the two days of study drug dosing.
26. Body mass index (BMI) great than 43.
27. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant. In some instances, patients whose medications or laboratory data meet exclusion criteria may participate at the Principal Investigator's discretion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Six-minute Walk Distance | Measured at baseline and 4 month follow-up
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin improves six-minute walk distance at 4-month follow-up

SECONDARY OUTCOMES:
Hand Grip Strength | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin improves hand grip strength at 4-month follow-up.
  readouts.
Short physical performance battery (SPPB) | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin improves the short physical performance battery (SPPB) at 4-month follow-up. SPPB range, range 0-12, 12-best
Number of cells with senescence markers | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin decreases cells with senescence markers in lower extremity adipose tissue, blood (CD3+ T lymphocytes), and gastrocnemius muscle at 4-month follow-up.
Gastrocnemius perfusion | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin improves gastrocnemius perfusion at 4-month follow-up. The investigators will use arterial spin labeling with magnetic resonance imaging (MRI) and post-cuff occlusion hyperemia to measure changes in calf perfusion at 3 Tesla. MRI perfusion will be measured using cuff occlusion hyperemia while the participant is supine. Gastrocnemius perfusion will be measured in ml/minute per 100g of tissue.

OTHER OUTCOMES:
Abundance of oxylipin dihomo-15d-PGJ2 | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin changes abundance of oxylipin dihomo-15d-PGJ2 in blood at 4-month follow-up.
Abundance of interleukin-6 markers | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin changes abundance of interleukin-6 (IL-6) markers in blood at 4-month follow-up. Quantitative reverse transcription-PCR (qRT-PCR) will be performed by Dr. Peterson's lab for RNA encoding IL-6 markers in adipose tissue, including interleukin-8 (IL-8), monocyte chemoattractant protein-1 (MCP-1), IL-1α, growth differentiation factor 15, and IL-6. Abundance of IL-6 markers will be measured in units of pg/mL.
Gastrocnemius muscle fibrosis | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether reduced senescent cell abundance and whether reduced IL-6 factor abundance in blood, gastrocnemius muscle, and adipose tissue, respectively, are correlated with reduced gastrocnemius muscle fibrosis at 4-month follow up. Antibodies to collagen I and III will quantify extracellular matrix composition. Picrosirius Red histochemistry will quantify total fibrous collagen, with polarized light to assess collagen organization.
Gastrocnemius muscle collagen | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether reduced senescent cell abundance and whether reduced IL-6 factor abundance in blood, gastrocnemius muscle, and adipose tissue, respectively, are correlated with reduced gastrocnemius muscle collagen at 4-month follow up. Antibodies to collagen I and III will quantify extracellular matrix composition. Picrosirius Red histochemistry will quantify total fibrous collagen, with polarized light to assess collagen organization.
Abundance of cells with increased myofiber size | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether reduced senescent cell abundance and whether reduced IL-6 factor abundance in blood, gastrocnemius muscle, and adipose tissue, respectively, are correlated with a reduced abundance of cells with increased myofiber size at 4-month follow up. Muscle fiber cross-sectional area will be quantified and 4',6-diamidino-2-phenylindole (DAPI) staining performed for centrally nucleated fibers, a marker of ischemic injury/regeneration.
Abundance of cells with central nuclei | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether reduced senescent cell abundance and whether reduced IL-6 factor abundance in blood, gastrocnemius muscle, and adipose tissue, respectively, are correlated with a reduced abundance of cells with central nuclei at 4-month follow up. Muscle fiber cross-sectional area will be quantified and DAPI staining performed for centrally nucleated fibers, a marker of ischemic injury/regeneration.
Interleukin-6 mRNA abundance | Measured at baseline and 4 months
  Among older people with PAD, the investigators will determine whether, compared to placebo, fisetin changes IL-6 mRNA abundance in gastrocnemius muscle and lower extremity adipose tissue at 4-month follow-up. qRT-PCR will quantify IL-6 mRNAs as described for fat tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States